CLINICAL TRIAL: NCT03804762
Title: Feasibility of the Third Space Robotic and Endoscopic Cooperative Surgery(TS-RECS) for Treating Gastric Stromal Tumor
Brief Title: A New Method: the Third Space Robotic and Endoscopic Cooperative Surgery (TS-RECS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2018LSK-168
Record Dates: First submitted 2018-12-23; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-04

CONDITIONS: Gastric Soft Tissue Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients received treatment of TS-RECS (Experimental)
  Interventions: Procedure: the third space robotic and endoscopic cooperative surgery

INTERVENTIONS:
Procedure: the third space robotic and endoscopic cooperative surgery — This technique combines the endoscopic techniques and the merits of Da Vinci surgical robot, such as flexible and precise instruments, tremors filtering system and a 3-D surgical view, and take full advantage of the methodology of the third space to dissect gastric submucosal tumors.

SUMMARY:
The third space robotic and endoscopic cooperative surgery (TS-RECS) combines the endoscopic techniques and the merits of Da Vinci surgical robot, such as flexible and precise instruments, tremors filtering system and a 3-D surgical view. TS-RECS takes full advantage of the methodology of the third space, making it possible to dissect gastric GISTs (gastrointestinal stromal tumors) entirely without the damage of mucosal layer. Here, this study preliminarily assessed the feasibility, safety and effectivity of the novel hybrid operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric GISTs originating from muscularis propria diagnosed by EUS (endoscopic ultrasound)；
* The maximal cross-sectional diameter of tumor ranging from 2cm to 5cm, or the maximal cross-sectional diameter of tumor <2cm but with malignant potential ( irregular shape, cystic space, heterogeneity and rapid growth during follow-ups ) ；
* No evidence of tumor metastasis on all per-operative evaluations；

Exclusion Criteria:

* 1. Patients with serious systemic comorbidities, such as severe heart failure, respiratory failure, uncontrolled hypertension;
* 2. Patients with advanced malignant tumor;
* 3. Patients were required the emergency operation by complete intestinal obstruction, perforation and hemorrhage caused by the tumor;
* 4.Patients with ulcer penetration into tumors;
* 5. Patients with the contraindications for general anesthesia;
* 6. Patients were pregnant or younger than 18 years old；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
the rate of adverse events | through study completion, an average of 6 months
  Adverse events included intraoperative adverse (full-thickness perforation, hemorrhage, injury of visceral organs and vessel, and anaesthesia complications), and postoperative adverse events (infectious complications, intra-abdominal /intraluminal bleeding, gastric stasis and leakage)

SECONDARY OUTCOMES:
rate of en bloc resection | 1 day
  the en bloc resection was defined as complete tumor resection with negative surgical margin.
the rate of intact mucosal layer | 1 day
  intact mucosal layer was defined as the tumor resection without full-thickness incision caused by operation
operation time | 1 day
  Operation time was defined from the time of docking to the time of trocar incision closure.
estimated blood loss | 1 day
  Blood loss was estimated through the analysis of the surgical and anaesthesiological reports.
time to oral diet | 30 days
  time to oral diet to assess the postoperative course.
duration of postoperative hospital stay | 30 days
  From the day of operation to the day of discharged, duration of postoperative hospital stay to assess the postoperative course.

CONTACTS AND LOCATIONS:
Overall Officials: Junjun She, MD,PHD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi F, Li Y, Pan Y, Sun Q, Wang G, Yu T, Shi C, Li Y, Xia H, She J. Clinical feasibility and safety of third space robotic and endoscopic cooperative surgery for gastric gastrointestinal stromal tumors dissection : A new surgical technique for treating gastric GISTs. Surg Endosc. 2019 Dec;33(12):4192-4200. doi: 10.1007/s00464-019-07223-w. Epub 2019 Oct 17. PMID 31624942